CLINICAL TRIAL: NCT06883500
Title: Design and Validation of an Energy Level Diary for Fatigue Management in Patients With Post-COVID Syndrome
Brief Title: Energy Level Diary for Patients With Post-COVID Syndrome
Status: Completed | Type: Observational
Sponsor: University of Witten/Herdecke (Other)
Responsible Party: Sponsor
Other Study IDs: PCS_EnergyDiary
Record Dates: First submitted 2025-03-18; First posted 2025-03-19 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: Post COVID Syndrome; Chronic Fatigue Symptoms
Keywords: post-covid syndrom; chronic fatigue syndrome; energy diary; rehabilitation
MeSH Terms: conditions — Fatigue Syndrome, Chronic

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients in neurological and cardiological rehablitation with Post-Covid Syndrome: A co-design approach was used and the diary was developed over three phases through repeated feedback loops including interviews with patients with PCS and an expert consensus, consisting of doctors, scientists, and therapists, using the Delphi method.
  Interventions: Behavioral: Energy diary

INTERVENTIONS:
Behavioral: Energy diary — A prospective observational study is conducted at two German rehabilitation centers in a co-design approach with repeated feedback loops (expert consensus, patient interviews). Daily energy-changes will be analyzed and validated using the Multidimensional Fatigue Inventory-20 (MFI-20).
  Other Names: MFI-20

SUMMARY:
Post-COVID-19 Syndrome (PCS) is characterized by symptoms, including fatigue, reduced physical performance, dyspnea, cognitive impairment, and psychological distress. Pateints have difficulties with energy management and often feel drained even after simple motor or cognitive tasks, which often leads to so called Crashes, after which patients are often bedridden for several day. This study examined wether an energy diary would facilitate the process of pacing during rehabilitation and beyond.

DETAILED DESCRIPTION:
Since the COVID-19 pandemic began, rehabilitation facilities have seen an influx of patients suffering from Post-COVID Syndrome (PCS), also referred to as postacute sequelae of SARS-CoV-2 infection (PASC).

PCS is characterized by symptoms persisting for more than 12 weeks post-infection, including chronic cognitive and motor fatigue, muscle pain, headaches, balance issues, autonomic dysfunction, sleep disturbances, and memory difficulties. Chronic fatigue syndrome (CFS), while lacking a universally accepted definition, can be understood as an intense fatigue that interferes with daily activities and worsens under stress. Patients often describe a significant lack of mental energy and muscle strength, with prolonged recovery times following physical exertion. The presence of Post-Exertional Malaise (PEM), which exacerbates symptoms after inadequate physical or mental activity, further complicates the clinical picture, causing overlap with symptoms of myalgic encephalomyelitis/chronic fatigue syndrome (ME/CFS).

The impact of PCS and chronic fatigue on patients' occupational, educational, and social activities can be as severe as that seen in other chronic illnesses, such as multiple sclerosis or cancer, leading to substantial economic burdens. Therefore, the demand for effective rehabilitation approaches is critical. However, managing fatigue presents challenges, as it may limit both the number and effectiveness of therapy sessions. It is essential to balance activity levels to prevent exacerbation of symptoms, making energy management a key component of therapeutic guidance.

The cognitive behavioral approach of "Pacing," which encourages patients to maintain a manageable level of activity without worsening symptoms, has been suggested for ME/CFS management. The PACE trial indicated that cognitive behavioral therapy and graded exercise therapy could support effective pacing, though these findings have sparked debate. A recent meta-analysis found that pacing interventions significantly reduced fatigue and psychosocial distress, particularly when participants were encouraged to gradually increase physical and cognitive activities. Nevertheless, there is a call for further randomized controlled trials (RCTs) using standardized pacing methods over longer durations, as current practices vary widely.

A retrospective analysis involving 86 PCS patients indicated that adherence to pacing, as measured by the Engagement in Pacing subscale (EPS), correlated with quicker recovery and symptom improvement. This aligns with recommendations to avoid both overexertion and underexertion in PCS cases. Consequently, graded exercise therapy may not be suitable in this context.

Diaries can serve as valuable tools for individuals to document their health experiences over time, revealing symptom and behavior trends with less recall bias compared to traditional questionnaires. In various medical fields, diaries have proven useful for evaluating behavior and therapy efficacy. With the rise of digital applications, tracking health behaviors has become more accessible, offering substantial data for analysis. However, a validated PCS-specific diary, created in collaboration with PCS patients, is currently lacking.

The present study aims to develop such a diary to monitor energy levels of patients with PCS throughout their rehabilitation process, hypothesizing that it will effectively document the impact of different therapies on daily energy levels.

ELIGIBILITY:
Inclusion Criteria:

history of (at least one) COVID-19 infection (positive PCR test at the time of infection), and ongoing or newly expressed performance deficits lasting for at least 3 months prior to recruitment.

Exclusion Criteria:

age below 18

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with PCS referred for medical rehabilitation at Clinic Koenigsfeld Ennepetal, Germany and Neurological Therapy Center Cologne, Germany
Sampling Method: Probability Sample
Enrollment: 66 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2024-04-01 (Actual); Study Completion 2024-09-30 (Actual)

PRIMARY OUTCOMES:
energy level according to energy diary | 2 years
  In an initial step, a diary was developed by experts together with patients (co-design). Versions of the diary were then provided to patients to investigate usability as well as sensitivity to daily changes in fatigue/ energy levels. Patient interviews were performed to collect feedback. The final version of the diary was validated against the Multidimensional Fatigue Inventory-20 (MFI-20). Patients completed the diary during inpatient (Koenigsfeld) and outpatient (Cologne) medical rehabilitation both including a combination of physical, cognitive and respiratory training as well as relaxation- and psychotherapy as indicated.

CONTACTS AND LOCATIONS:
Locations (2):
- Germany (2):
  - Neurologic Therapy Center Cologne, Cologne, North Rhine-Westphalia
  - Clinic Königsfeld,, Ennepetal, North Rhine-Westphalia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Balke M, Garbsch R, Cormann J, Pape P, Mooren FC, Schmitz B. Design and validation of an energy level diary for fatigue management in patients with post-COVID syndrome. Front Rehabil Sci. 2025 Jul 21;6:1633466. doi: 10.3389/fresc.2025.1633466. eCollection 2025. PMID 40761505